CLINICAL TRIAL: NCT02884739
Title: The Mortality and Its Associated Factors in Schizophrenia Patients Older Than 60 Years
Brief Title: Mental Healthcare in Older Adults With Schizophrenia
Acronym: CSA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PN08001
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Schizophrenia; Chronic Psychiatric Disorder
MeSH Terms: conditions — Schizophrenia | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- schizophrenia
  Interventions: Other: Data collection
- chronic psychiatric disorder other than schizophrenia
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection

SUMMARY:
As in the general population, there is a gradual and steady increase in life expectancy of patients with schizophrenia. But this increase is at a smaller scale, with a rate of premature death that is still 2 to 3 times higher than that found in the general population. This excessive early mortality is explained by an overrepresentation of suicide deaths, but also a higher prevalence of somatic diseases, mainly cardiovascular. But today there are only very few epidemiological data on the mortality of patients with schizophrenia, including those aged over 60 years. What are the sociodemographic and clinical characteristics (psychiatric and somatic) of these schizophrenic elderly patients? Do they benefit from a somatic follow-up adequate and systematic? What are their levels of social independence and of quality of life? the answers these questions and the description of the offer of geriatric care and of psychiatric care currently provided by different sectors of psychiatry in France is an indispensable prerequisite for any project to improve the quality of life, state of health and mortality of older patients with schizophrenia.

DETAILED DESCRIPTION:
Evaluate prospectively over 5 years, the rates and causes of mortality in a cohort of schizophrenic patients older than 60 years, followed by adult psychiatry sectors, compared to those patients matched for sex and age and monitored by the same sectors for a chronic psychiatric disorder other than schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged than 60 years with a diagnosis of schizophrenia, according to the DSM-IV criteria
* Men or women aged than 60 years with chronic psychiatric disorder other than schizophrenia
* Patients consenting to participate to the study
* Patients enrolled in the national healthcare insurance program

Exclusion Criteria:

-Disease affecting the central nervous system

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia and patients with chronic psychiatric disorder other than schizophrenia were included
Sampling Method: Non-Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2010-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Death | 5 years
  Death of any causes

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Raucher-Chene D, Hoertel N, Bera-Potelle C, Terrien S, Barriere S, Da Rin D, Tran E, Cuervo-Lombard C, Portefaix C, Limosin F. Mental healthcare in older adults with schizophrenia: results from 118 French public psychiatric departments. Int Psychogeriatr. 2015 Oct;27(10):1749-50. doi: 10.1017/S1041610215001064. Epub 2015 Jul 6. No abstract available. PMID 26144544